CLINICAL TRIAL: NCT05505032
Title: Optimal FiO2 Value, Oxygen Reserve Index, and Prevention of Hyperoxemia in Children: A Prospective, Randomized, Single-blind Study
Brief Title: Oxygen Reserve Index and Prevention of Hyperoxemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Uslu, Principal Investigator, Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-05/1838
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Hyperoxemia; Oxygen Reserve Index; Hyperoxia; Fraction of Inspired Oxygen
Keywords: Oxygen Reserve Index; Hyperoxemia; Hyperoxia; Fraction of Inspired Oxygen
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Group F30 : FiO2 value is %30 Group F50 : FiO2 value is %50 Group F80 : FiO2 value is %80
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group F30 (Experimental): In these patients, the FiO2 value will be adjusted to 30% in the perioperative period.
  Interventions: Drug: Oxygen; Device: Masimo Root Radical 7
- Group F50 (Experimental): In these patients, the FiO2 value will be adjusted to 50% in the perioperative period.
  Interventions: Drug: Oxygen; Device: Masimo Root Radical 7
- Group F80 (Experimental): In these patients, the FiO2 value will be adjusted to 80% in the perioperative period.
  Interventions: Drug: Oxygen; Device: Masimo Root Radical 7

INTERVENTIONS:
Drug: Oxygen — Determination of FiO2 threshold value as an indicator of hyperoxemia in anesthesia stages.
Device: Masimo Root Radical 7 — We use it to measure the oxygen reserve index (ORi).

SUMMARY:
In patients under general anesthesia, the oxygen level (FiO2) used in inspiration is usually adjusted by monitoring the peripheral oxygen saturation level (SpO2). As a non-invasive method, SpO2 monitoring is known as one of the required methods that can be used to adjust FiO2 and detect and treat hypoxemia. While SpO2 approaching 100% matches the value of 128 mmHg in arterial partial oxygen pressure (PaO2), in cases where PaO2 increases more, the investigators cannot follow this situation with SpO2 and cannot prevent hyperoxemia.

As stated in the literature, hyperoxemia has positive effects in general anesthesia and intensive care, as well as negative effects such as increased inflammation, oxidative stress and ischemia-reperfusion. In addition, acute lung injury, development of atelectasis, increased mortality, and critical illness rates have been associated with hyperoxemia in many publications. The only way the investigators can use to measure the level of hyperoxemia seems to be arterial blood gas analysis, and this method limits the investigators use because it is invasive. The Oxygen Reserve Index (ORi™) (Masimo Corp., Irvine, CA, USA) is a variable related to real-time oxygenation reserve status in the mildly hyperoxemic range (approximately 100 - 200 mmHg PaO2). ORi can be defined as a multi-wavelength, noninvasive pulse co-oximetry sensor. ORi is a dimensionless index ranging from 0.00 (no reserve) to 1.00 (maximum reserve) depending on the oxygenation reserve status.

There are very few studies in the literature using ORi to detect hyperoxemia. The investigators thought that if FiO2 levels used in preoxygenation, anesthesia maintenance and recovery stages in day surgeries were correlated with ORi levels, a threshold value could be determined for FiO2 levels during anesthesia stages in cases where invasive arterial blood gas could not be followed.

This study aims to determine the relationship between SpO2, FiO2 and ORi during general anesthesia, to investigate the usefulness of ORi in determining the FiO2 threshold value during anesthesia stages as an indicator of hyperoxemia, and to investigate the effects of these values on the hemodynamics, recovery, agitation and nausea-vomiting states of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an American Society of Anesthesiologists (ASA) score of 1

Exclusion Criteria:

* Patients with an American Society of Anesthesiologists (ASA) score of 2 and above

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
FiO2 threshold value | Until the surgery is over
  Correlation of FiO2 threshold value and ORi value

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided